CLINICAL TRIAL: NCT00002865
Title: HIGH INTENSITY, BRIEF DURATION CHEMOTHERAPY FOR RELAPSED OR REFRACTORY ALL: A PHASE II STUDY OF A MULTIDRUG REGIMEN
Brief Title: High-Intensity, Brief-Duration Chemotherapy in Treating Patients With Relapsed or Refractory Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065137; CCCWFU-21195; NCI-V96-1062
Record Dates: First submitted 1999-11-01; First posted 2004-08-11 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Leukemia
Keywords: recurrent adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Etoposide; Ifosfamide; Leucovorin; Mesna; Methotrexate; Hydrocortisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: leucovorin calcium
Drug: mesna
Drug: methotrexate
Drug: therapeutic hydrocortisone
Drug: vincristine sulfate
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of high-intensity, brief-duration chemotherapy in treating patients with relapsed or refractory acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete response rate to high-intensity, brief-duration chemotherapy with cyclophosphamide, methotrexate, vincristine, doxorubicin, and dexamethasone followed by ifosfamide, methotrexate, vincristine, cytarabine, etoposide, and dexamethasone in patients with relapsed or refractory acute lymphocytic leukemia (ALL). II. Determine the toxic effects of these regimens in these patients.

OUTLINE: All patients receive up to six alternating courses (every 3-4 weeks) of two chemotherapy regimens: cyclophosphamide, oral dexamethasone, methotrexate with leucovorin rescue, vincristine, and doxorubicin over 5 days; and ifosfamide/mesna, oral dexamethasone, methotrexate with leucovorin rescue, vincristine, cytarabine, and etoposide over 5 days. G-CSF is given following each course until recovery of the neutrophil count. All patients receive triple intrathecal chemotherapy on day 1. Patients with CNS disease receive intrathecal therapy twice weekly until the CSF is clear, then weekly for 4 weeks, and monthly for 1 year; those who have not received prior CNS irradiation also receive whole-brain radiotherapy. Patients are followed monthly for 6 months, every 3 months for 18 months, every 6 months for 2 years, then annually.

PROJECTED ACCRUAL: A total of 37 evaluable patients will be accrued if at least 4 of the first 17 patients respond.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed acute lymphocytic leukemia that is relapsed after or refractory to induction therapy 1 or 2 prior inductions allowed, but refractory to only 1 regimen CNS involvement allowed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: 0-3 Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 times normal (unless directly attributable to leukemia) Renal: Creatinine no greater than 1.5 times normal (unless directly attributable to leukemia) Cardiovascular: No uncontrolled or severe cardiovascular disease including: Myocardial infarction within 6 months Congestive heart failure Other: No uncontrolled duodenal ulcer No uncontrolled infection No second malignancy within 5 years except curatively treated: In situ cervical cancer Basal cell skin cancer No other serious medical illness that would limit survival to under 2 years No psychiatric illness that would prevent informed consent or compliance No pregnant or nursing women Adequate contraception required of fertile patients

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1995-04; Primary Completion 2000-06 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
response rate for patients with relapsed or refractory acute lymphoblastic leukemia after brief, high intensity chemotherapy | 14 days
evaluate adverse events after brief, high intensity chemotherapy | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayard L. Powell, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States